CLINICAL TRIAL: NCT04892446
Title: A Phase 2 Multi-Arm Study of Magrolimab Combinations in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Study of Magrolimab Combinations in Patients With Relapsed/Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated early due to the Sponsor's decision to discontinue development of the investigational drug and close the program.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-558-5915; 2021-001798-21 (EudraCT Number)
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Results first posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — magrolimab; daratumumab; pomalidomide; Dexamethasone; Bortezomib; carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Magrolimab+Daratumumab (Experimental): Participants with relapsed/refractory multiple myeloma (MM) who have had 3 or more prior therapies including an immunomodulatory drug (IMiD) and a proteasome inhibitor (PI) will receive magrolimab as per protocol and daratumumab 1800 mg subcutaneously (SC) or 16 milligrams per kilogram (mg/kg) intravenously (IV) on Days 8, 15, 22, 29 of Cycle 1, Days 1, 8, 15, 22 of Cycle 2 and Days 1 and 15 (every 2 weeks) until Cycle 6 (total of 8 doses) followed by Day 1 (every 4 weeks) for subsequent cycles. (Cycle 1=35 days, All other Cycles=28 days).
  Interventions: Drug: Magrolimab; Drug: Daratumumab
- Magrolimab+Pomalidomide+Dexamethasone (Experimental): Participants with relapsed/refractory multiple myeloma who have had 3 or more prior therapies including an IMiD and a PI will receive magrolimab as per protocol and pomalidomide 4 mg on Days 1 to 21 (daily) of Cycle 1, Days 1 to 21 (daily) of Cycle 2 and onward and dexamethasone 40 mg on Days 1, 8, 15, 22, 29 of Cycle 1, Days 1, 8, 15, 22 of Cycle 2 and onward. (Cycle 1=35 days, All other Cycles=28 days).
  Interventions: Drug: Magrolimab; Drug: Pomalidomide; Drug: Dexamethasone
- Magrolimab+Carfilzomib+Dexamethasone (Experimental): Participants with relapsed/refractory multiple myeloma who have had 3 or more prior therapies including an IMiD and a PI will receive magrolimab as per protocol and carfilzomib 20 mg/m^2 on Days 8, 15, 22 of Cycle 1, Days 1, 8, 15 of Cycle 2 and onward (if the carfilzomib starting dose of 20 mg/m^2 is tolerated after Cycle 1, Day 8, the dose will be escalated to 70 mg/m^2 on Cycle 1, Day 15 and thereafter) and dexamethasone 40 mg on Days 1, 8, 15, 22, 29 of Cycle 1, Days 1, 8, 15, 22 of Cycles 2 to 9 and then Days 1, 8, 15 from Cycle 10 and onward. (Cycle 1=35 days, All other Cycles=28 days).
  Interventions: Drug: Magrolimab; Drug: Dexamethasone; Drug: Carfilzomib
- Magrolimab+Bortezomib+Dexamethasone (Experimental): Bortezomib + Dexamethasone may be initiated based on the preliminary safety and efficacy of the Carfilzomib + Dexamethasone cohort.
  Participants with relapsed/refractory multiple myeloma who have had 1 or more prior therapies including an IMiD and a PI will receive magrolimab as per protocol and carfilzomib 1.3 mg/m^2 on Days 8, 15, 22, 29 of Cycle 1, Days 1, 8, 15, 22 of Cycle 2 and onward (Maximum of 8 cycles in those who have previously received bortezomib) and dexamethasone 40 mg on Days 1, 8, 15, 22, 29 of Cycle 1, Days 1, 8, 15, 22 of Cycles 2 to 9 and then Days 1, 8, and 15 from Cycle 10 and onward. (Cycle 1=35 days, All other Cycles=28 days).
  Interventions: Drug: Magrolimab; Drug: Dexamethasone; Drug: Bortezomib

INTERVENTIONS:
Drug: Magrolimab — Administered IV
  Other Names: GS-4721
Drug: Daratumumab — Administered either SC or IV
  Arms: Magrolimab+Daratumumab
Drug: Pomalidomide — Administered orally
  Arms: Magrolimab+Pomalidomide+Dexamethasone
Drug: Dexamethasone — Administered orally
  Arms: Magrolimab+Bortezomib+Dexamethasone; Magrolimab+Carfilzomib+Dexamethasone; Magrolimab+Pomalidomide+Dexamethasone
Drug: Bortezomib — Administered either SC or IV
  Arms: Magrolimab+Bortezomib+Dexamethasone
Drug: Carfilzomib — Administered IV
  Arms: Magrolimab+Carfilzomib+Dexamethasone

SUMMARY:
The goal of this clinical study is to learn more about the safety and dosing of the study drug, magrolimab, in combination with other anticancer therapies in participants with relapsed/refractory multiple myeloma.

ELIGIBILITY:
Key Inclusion Criteria:

All Individuals:

* Have been previously diagnosed with MM based on the International Myeloma Working Group (IMWG) 2016 criteria and currently requires treatment.
* Must have measurable disease as defined by 1 or more of the following:

  * Serum monoclonal protein (M-protein) ≥ 0.5 grams per deciliter (g/dL) (greater than or equal to [≥] 5 grams per liter [g/L]).
  * Urine M-protein ≥ 200 mg/24 hours (h).
  * Serum free light chain (SFLC) assay: involved SFLC level ≥ 10 mg/dL (100 mg/L) with abnormal SFLC ratio.
* Has provided informed consent.
* Is willing and able to comply with clinic visits and procedure outlined in the study protocol.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Life expectancy ≥ 3 months.
* Absolute neutrophil count (ANC) ≥ 1000 cells/uL (1.0 x 10^9/L); granulocyte colony-stimulating factor (G-CSF) is not permitted within 1 week of screening to meet eligibility criteria.
* Platelet count ≥ 75,000 cells/uL (75 x 10^9/L); platelet transfusion is not permitted within 1 week of screening to meet eligibility criteria.
* Hemoglobin ≥ 9 g/dL; prior to initial dose of study treatment. Note: Transfusions are allowed to meet hemoglobin eligibility
* Adequate liver function as demonstrated by the following:

  * Aspartate aminotransferase (AST) ≤ 3.0 x upper limit of normal (ULN).
  * Alanine aminotransferase (ALT) ≤ 3.0 x ULN.
  * Total bilirubin ≤ 1.5 x ULN (or ≤ 3.0 x ULN and primarily unconjugated if individual has a documented history of Gilbert's syndrome or genetic equivalent).
* International normalized ratio (INR) ≤ 1.2; Individuals receiving anticoagulation treatment may be allowed to participate if INR is within the therapeutic range prior to alternate assignment.
* Individuals must have adequate renal function as demonstrated by a creatinine clearance ≥ 30 mL/min calculated by the Cockcroft-Gault formula or measured by 24 hours urine collection.
* Corrected serum calcium ≤ 2.9 millimoles per liter (mmol/L) (11.5 mg/dL); measures to reduce calcium to acceptable levels, such as a short course of steroids, bisphosphonates, hydration, or calcitonin are acceptable.
* Pretreatment blood cross-match completed.
* Males and females of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception.
* Must be willing to consent to mandatory pretreatment and on-treatment bone marrow biopsies (trephines).
* Magrolimab in Combination with Daratumumab: In addition to fulfilling the inclusion criteria for all individuals, individuals who are assigned to receive magrolimab in combination with daratumumab should fulfill the following:

  * Must have received at least 3 previous lines of therapy for MM including an IMiD such as lenalidomide and a PI such as bortezomib.
  * Individuals must have not had prior anti-cluster differentiation 38 (CD38) antibody therapy for at least 6 months prior to enrollment.
  * No prior history of discontinuation of daratumumab due to toxicity.
* Magrolimab in Combination with Pomalidomide and Dexamethasone: In addition to fulfilling the inclusion criteria for all Individuals, Individuals who are assigned to receive magrolimab in combination with pomalidomide and dexamethasone should fulfill the following:

  * Must have received at least 3 previous lines of therapy for MM including an IMiD such as lenalidomide and a PI such as bortezomib.
  * Prior treatment with pomalidomide is allowed if the Individual achieved at least a partial response (PR) to the most recent pomalidomide therapy and will have had at least a 6-month treatment-free interval from the last dose of pomalidomide until first study treatment.
  * No prior history of discontinuation of pomalidomide due to toxicity.
  * No contraindication to dexamethasone.
* Magrolimab in Combination with Carfilzomib and Dexamethasone: In addition to fulfilling the inclusion criteria for all patients, patients who are assigned to receive magrolimab in combination with carfilzomib and dexamethasone should fulfill the following:

  * Patient must have received at least 3 previous lines of therapy for MM including an IMiD such as lenalidomide and a PI such as bortezomib.
  * Prior treatment with a PI, including carfilzomib, is allowed if the patient achieved at least a PR to the most recent prior PI therapy, and will have had at least a 6-month PI treatment-free interval from the last dose until first study treatment.
  * No prior history of discontinuation of carfilzomib due to toxicity.
  * No contraindication to dexamethasone
* Magrolimab in Combination with Bortezomib and Dexamethasone: In addition to fulfilling the inclusion criteria for all individuals, individuals who are assigned to receive magrolimab in combination with bortezomib and dexamethasone should fulfill the following:

  * Must have received at least 1 previous line of therapy for MM including an IMiD such as lenalidomide and a PI such as bortezomib.
  * Prior treatment with a PI, including bortezomib, is allowed if the Individual achieved at least a PR to the most recent prior PI therapy, and will have had at least a 6-month PI treatment-free interval from the last dose until first study treatment.
  * No prior history of discontinuation of bortezomib due to toxicity.
  * No contraindication to dexamethasone.

Key Exclusion Criteria:

* Individuals with known amyloidosis including myeloma complicated by amyloidosis.
* Multiple myeloma of immunoglobulin M subtype.
* Individuals with Waldenstrom's macroglobulinemia.
* Individuals with myelodysplastic syndrome (MDS).
* Plasma cell leukemia (defined as either 20% of peripheral blood white blood cell (WBC) count comprised of plasma/CD138-positive cells) or circulating plasma cells ≥ 2 x 10^9/L.
* Individuals with solitary bone or extramedullary plasmacytoma as the only evidence of plasma cell dyscrasia.
* Polyneuropathy, Organomegaly, Endocrinopathy, Monoclonal protein, Skin changes (POEMS) syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, M-protein, and skin changes).
* Glucocorticoid therapy (prednisone > 40 mg/day or equivalent) within 14 days prior to enrollment; corticosteroid therapy for hypercalcemia is allowed.
* Chemotherapy with approved or investigational anticancer therapeutics within 28 days prior to enrollment.
* Focal radiation therapy within 7 days prior to enrollment; radiation therapy to an extended field involving a significant volume of bone marrow within 21 days prior to enrollment (ie, prior radiation must have been to less than 30% of the bone marrow).
* Immunotherapy within 28 days prior to enrollment.
* Major surgery (excluding procedures to stabilize the vertebrae) within 28 days prior to enrollment.
* Positive serum pregnancy test.
* Breastfeeding female.
* Known hypersensitivity to any of the study drugs, the metabolites, or formulation excipient.
* Prior treatment with CD47 or signal regulatory protein alpha (SIRPα)-targeting agents.
* Current participation in another interventional clinical trial.
* Autologous stem cell transplant < 100 days prior to enrollment.
* Considered eligible to receive autologous or allogeneic stem cell transplant (SCT) at the time of enrollment.
* Allogeneic SCT for the treatment of MM within 6 months of enrollment or active graft-versus-host disease requiring immunosuppression.
* Significant neuropathy (Grade 3 to 4, or Grade 2 with pain) within 14 days prior to enrollment.
* Known inherited or acquired bleeding disorders.
* Known cirrhosis.
* Clinical suspicion or documentation of central nervous system (CNS) disease.
* Significant disease or medical conditions, as assessed by the investigator and sponsor, that would substantially increase the risk-benefit ratio of participating in the study. This includes, but is not limited to, acute myocardial infarction within the last 6 months, unstable angina, uncontrolled diabetes mellitus, significant active infections, congestive heart failure, or New York Heart Association (NYHA) Class III or IV heart failure.
* Acute active infection requiring systemic antibiotics, antiviral (except antiviral therapy directed against reactivation) or antifungal agents within 14 days prior to enrollment.
* Second malignancy, except treated basal cell or localized squamous skin carcinomas, localized prostate cancer, or other malignancies for which patients are not on active anticancer therapies and have had no evidence of active malignancy for at least 1 year. Other exceptions may be considered with sponsor approval. Previous hormonal therapy with luteinizing hormone-releasing hormone agonists for prostate cancer and treatment with bisphosphonates and receptor activator of nuclear factor kappa-B ligand (RANKL) inhibitors are not criteria for exclusion.
* Known active or chronic hepatitis B or C infection or human immunodeficiency virus (HIV) infection in medical history.
* Active hepatitis B virus (HBV) and/or active hepatitis C virus (HCV), and/or HIV infection following testing at screening:
* Individuals who test positive for hepatitis B surface antigen (HBsAg). Patients who test positive for hepatitis B core antibody (anti-HBc) will require HBV DNA by quantitative polymerase chain reaction (PCR) for confirmation of active disease.
* Individuals who test positive for HCV antibody. Patients who test positive for HCV antibody will require HCV ribonucleic acid (RNA) by quantitative PCR for confirmation of active disease.
* Individuals who test positive for HIV.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (22):
- United States (16):
  - Arizona Oncology Associates , PC - HOPE, Tucson, Arizona
  - US San Diego Moores Cancer Center, La Jolla, California
  - Stanford Cancer Institute, Palo Alto, California
  - Karmanos Cancer Institute, Detroit, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center - Main Campus, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Cleveland Clinic - Taussig Cancer Institute, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Bend Memorial Clinic, P.C. d/b/a Summit Health, Bend, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - US Oncology, Inc. IRB, Dallas, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - US Oncology, Inc., IRB, Fairfax, Virginia
- Canada (2):
  - Cross Cancer Institute, Edmonton
  - Princess Margaret Cancer Centre, Toronto
- Czechia (4):
  - Fakultní nemocnice Brno, Brno
  - Fakultní Nemocnice Olomouc, Olomouc
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Fakultní nemocnice Ostrava, Severomoravsky KRAJ

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paul B, Liedtke M, Khouri J, Rifkin R, Gandhi MD, Kin A, Levy MY, Silbermann R, Cottini F, Sborov DW, Sandhu I, Villarreal L, Murphy M, Gu L, Chen A, Rajakumaraswamy N, Usmani SZ. A phase II multi-arm study of magrolimab combinations in patients with relapsed/refractory multiple myeloma. Future Oncol. 2023 Jan;19(1):7-17. doi: 10.2217/fon-2022-0975. Epub 2023 Feb 13. PMID 36779512
- [Background] Paul B, Minarik J, Cottini F, Gasparetto C, Khouri J, Gandhi M, et al. Safety and Tolerability of Magrolimab Combinations in Patients With Relapsed/Refractory Multiple Myeloma: Safety Run-in Results From a Phase 2 Study [Poster 3383]. 65th American Society of Hematology (ASH) Annual Meeting; 2023 December 9-12; San Diego, California.
- [Derived] Paul B, Minarik J, Cottini F, Gasparetto C, Khouri J, Gandhi M, Hillengass J, Levy M, Liedtke M, Manda S, Sandhu I, Sborov D, Spicka I, Usmani S, Dong M, Gu L, Leung C, Doshi P, Chen C, Pour L. Final Results of a Phase 2 Multi-Arm Study of Magrolimab Combinations in Patients With Relapsed/Refractory Multiple Myeloma. EJHaem. 2025 Jun 6;6(3):e70072. doi: 10.1002/jha2.70072. eCollection 2025 Jun. PMID 40485906
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-558-5915

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 43 participants were screened.
Pre-assignment Details: Participants were enrolled at study sites in the United States, Czech Republic, and Canada.
  Magrolimab in combination with bortezomib and dexamethasone cohort was not initiated due to early closure of study.
  As all participants were dosed with same dose of magrolimab, per prespecified analysis, data for Safety Run-in and corresponding Dose-expansion cohorts were combined except for dose limiting toxicity outcome measure, for which data was collected only in Safety Run-in Cohorts.
Groups:
- Magrolimab+Daratumumab: Participants in Safety Run-in and Dose-expansion period with relapsed/refractory multiple myeloma who have had 3 or more prior therapies including an immunomodulatory drug (IMiD) and a proteasome inhibitor (PI) received magrolimab intravenously (IV) 1 milligrams per kilogram (mg/kg) on Day 1 and 30 mg/kg on Days 8, 15, 22, 29 of Cycle 1; 30 mg/kg every week on Days 1, 8, 15, 22 of Cycle 2; 30 mg/kg on Days 1, 15 from Cycle 3 onwards.
  Participants also received daratumumab 1800 mg subcutaneously (SC) or 16 mg/kg IV on Days 8, 15, 22, 29 of Cycle 1; Days 1, 8, 15, 22 of Cycle 2; and Days 1, 15 (every 2 weeks) until Cycle 6 (total of 8 doses) followed by Day 1 (every 4 weeks) for subsequent cycles. (Cycle 1=35 days, All other Cycles=28 days).
- Magrolimab+Pomalidomide+Dexamethasone: Participants in Safety Run-in and Dose-expansion period with relapsed/refractory multiple myeloma who have had 3 or more prior therapies including an IMiD and a PI received magrolimab IV 1 mg/kg on Day 1 and 30 mg/kg on Days 8, 15, 22, 29 of Cycle 1; 30 mg/kg every week on Days 1, 8, 15, 22 of Cycle 2; 30 mg/kg on Days 1, 15 from Cycle 3 onwards.
  Participants also received pomalidomide orally 4 mg on Days 1 to 21 (daily) of Cycle 1 and onward and dexamethasone orally 40 mg on Days 1, 8, 15, 22, 29 of Cycle 1; Days 1, 8, 15, 22 of Cycle 2 and onward. (Cycle 1=35 days, All other Cycles=28 days).
- Magrolimab+Carfilzomib+Dexamethasone: Participants in Safety Run-in and Dose-expansion period with relapsed/refractory multiple myeloma who have had 3 or more prior therapies including an IMiD and a PI received magrolimab IV 1 mg/kg on Day 1 and 30 mg/kg on Days 8, 15, 22, 29 of Cycle 1; 30 mg/kg every week on Days 1, 8, 15, 22 of Cycle 2; 30 mg/kg on Days 1, 15 from Cycle 3 onwards.
  Participants also received carfilzomib IV 20 milligrams per square meter (mg/m^2) on Days 8, 15, 22 of Cycle 1; Days 1, 8, 15 of Cycle 2 and onward (if the carfilzomib starting dose of 20 mg/m^2 was tolerated after Cycle 1, Day 8, the dose was escalated to 70 mg/m^2 on Cycle 1, Day 15 and thereafter) and dexamethasone orally or IV 40 mg on Days 8, 15, 22, 29 of Cycle 1; Days 1, 8, 15, 22 of Cycles 2 to 9 and then Days 1, 8, 15 from Cycle 10 and onward. (Cycle 1=35 days, All other Cycles=28 days).
Period: Overall Study
Arm/Group | Magrolimab+Daratumumab | Magrolimab+Pomalidomide+Dexamethasone | Magrolimab+Carfilzomib+Dexamethasone
Started | 15 | 10 | 11
Completed | 7 | 5 | 8
Not Completed | 8 | 5 | 3
Not completed — Death | 4 | 4 | 0
Not completed — Withdrew consent | 3 | 0 | 1
Not completed — Investigator's discretion | 1 | 1 | 0
Not completed — Study terminated by sponsor | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who received at least 1 dose of study treatment with treatment group designated according to the actual treatment received.
  As all participants were dosed with same dose of magrolimab, per prespecified analysis, data for Safety Run-in and corresponding Dose-expansion cohorts were combined for all 3 arms.
Groups:
- Magrolimab+Daratumumab: Participants in Safety Run-in and Dose-expansion period with relapsed/refractory multiple myeloma who have had 3 or more prior therapies including an IMiD and a PI received magrolimab IV 1 mg/kg on Day 1 and 30 mg/kg on Days 8, 15, 22, 29 of Cycle 1; 30 mg/kg every week on Days 1, 8, 15, 22 of Cycle 2; 30 mg/kg on Days 1, 15 from Cycle 3 onwards.
  Participants also received daratumumab 1800 mg SC or 16 mg/kg IV on Days 8, 15, 22, 29 of Cycle 1; Days 1, 8, 15, 22 of Cycle 2; and Days 1, 15 (every 2 weeks) until Cycle 6 (total of 8 doses) followed by Day 1 (every 4 weeks) for subsequent cycles. (Cycle 1=35 days, All other Cycles=28 days).
- Magrolimab+Carfilzomib+Dexamethasone: Participants in Safety Run-in and Dose-expansion period with relapsed/refractory multiple myeloma who have had 3 or more prior therapies including an IMiD and a PI received magrolimab IV 1 mg/kg on Day 1 and 30 mg/kg on Days 8, 15, 22, 29 of Cycle 1; 30 mg/kg every week on Days 1, 8, 15, 22 of Cycle 2; 30 mg/kg on Days 1, 15 from Cycle 3 onwards.
  Participants also received carfilzomib IV 20 mg/m^2 on Days 8, 15, 22 of Cycle 1; Days 1, 8, 15 of Cycle 2 and onward (if the carfilzomib starting dose of 20 mg/m^2 was tolerated after Cycle 1, Day 8, the dose was escalated to 70 mg/m^2 on Cycle 1, Day 15 and thereafter) and dexamethasone orally or IV 40 mg on Days 8, 15, 22, 29 of Cycle 1; Days 1, 8, 15, 22 of Cycles 2 to 9 and then Days 1, 8, 15 from Cycle 10 and onward. (Cycle 1=35 days, All other Cycles=28 days).
- Total: Total of all reporting groups
Arm/Group | Magrolimab+Daratumumab | Magrolimab+Pomalidomide+Dexamethasone | Magrolimab+Carfilzomib+Dexamethasone | Total
Number analyzed (Participants) | 14 | 10 | 11 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 4 | 5 | 16
  >=65 years | 7 | 6 | 6 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (9.5) | 66 (10.2) | 68 (8.0) | 66 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 2 | 5 | 17
  Male | 4 | 8 | 6 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 10 | 11 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 1 | 1 | 1 | 3
  White | 11 | 9 | 10 | 30
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 2 | 1 | 4 | 7
  United States | 10 | 5 | 4 | 19
  Czechia | 2 | 4 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Dose-limiting Toxicities (DLTs) According to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Description: A DLT was defined as any Grade 3 or higher hematologic toxicity or Grade 3 or higher nonhematologic toxicity, that had worsened in severity from pretreatment baseline during the DLT assessment period and, in the opinion of the investigator, the adverse event (AE) was at least possibly related to magrolimab.
  Percentages are rounded off.
Time Frame: Up to 35 days
Population: The DLT-Evaluable Analysis Set included all participants in the Safety Analysis Set who were enrolled in the Safety Run-in cohorts and fulfilled the criteria for evaluation for DLT specified in the protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Magrolimab+Daratumumab | Magrolimab+Pomalidomide+Dexamethasone | Magrolimab+Carfilzomib+Dexamethasone
Number analyzed (Participants) | 6 | 6 | 6
percentage of participants | 16.7 | 16.7 | 0

2. Primary Outcome: Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAE's) According to the NCI CTCAE Version 5.0
Description: An AE is any untoward medical occurrence in a clinical study participant administered a study drug that does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of a study drug, whether or not the AE is considered related to the study drug. A treatment-emergent AE was defined as any AE that began on or after the date of first dose of any study drug up to the date of last dose of any study drug plus 70 days.
Time Frame: Up to 1.3 years plus 70 days
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Magrolimab+Daratumumab | Magrolimab+Pomalidomide+Dexamethasone | Magrolimab+Carfilzomib+Dexamethasone
Number analyzed (Participants) | 14 | 10 | 11
percentage of participants | 100 | 100 | 100

3. Primary Outcome: Percentage of Participants Experiencing Treatment-emergent Laboratory Abnormalities According to the NCI CTCAE Version 5.0
Description: Treatment-emergent laboratory abnormalities were defined as values that increase at least 1 toxicity grade from baseline at any postbaseline time point, up to and included the date of last dose of study drug plus 70 days for participants who permanently discontinued study drug, or the day before initiation of new anticancer therapy including stem cell transplant (SCT) (whichever was earlier). If the relevant baseline laboratory value was missing, any abnormality of at least Grade 1 observed within the time frame specified above was considered treatment emergent.
  Percentages are rounded off.
Time Frame: Up to 1.3 years plus 70 days
Population: Participants in the Safety Analysis Set were analyzed. As all participants were dosed with same dose of magrolimab, per prespecified analysis, data for Safety Run-in and corresponding Dose-expansion cohorts were combined for all 3 arms.
Measure: Number; unit: percentage of participants
Arm/Group | Magrolimab+Daratumumab | Magrolimab+Pomalidomide+Dexamethasone | Magrolimab+Carfilzomib+Dexamethasone
Number analyzed (Participants) | 14 | 10 | 11
percentage of participants
  Hematology: Any Grade 1 or Higher | 92.9 | 100 | 100
  Chemistry: Any Grade 1 or Higher | 92.9 | 100 | 100

4. Primary Outcome: Objective Response Rate (ORR)
Description: Objective response rate is defined as the percentage of participants who achieve confirmed stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR), as assessed by the investigator per the International Myeloma Working Group (IMWG) 2016 criteria. CR defined as negative immunofixation on serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow (BM) aspirates; sCR defined as CR as above plus normal serum free light-chain (FLC) assay ratio and absence of clonal cells in BM biopsy by immunohistochemistry; VGPR defined as serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥ 90% reduction in serum M-protein plus urine M-protein <100 mg/24 h; PR defined as ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 h.
  Percentages are rounded off.
Time Frame: Up to 1.5 years
Population: The Full Analysis Set included all participants who took ≥ 1 dose of study drugs with arm designated according to the planned treatment at enrollment.
  As all participants were dosed with same dose of magrolimab, per prespecified analysis, data for Safety Run-in and corresponding Dose-expansion cohorts were combined for all 3 arms.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Magrolimab+Daratumumab | Magrolimab+Pomalidomide+Dexamethasone | Magrolimab+Carfilzomib+Dexamethasone
Number analyzed (Participants) | 14 | 10 | 11
percentage of participants | 14.3 [1.8 to 42.8] | 20.0 [2.5 to 55.6] | 36.4 [10.9 to 69.2]

5. Secondary Outcome: Duration of Response (DoR)
Description: DoR was measured from earliest date of sCR, CR, VGPR, or PR, whichever was first recorded, until earliest date of documented progression disease (PD) per IMWG 2016, documented relapse, or death from any cause, whichever occurred first. sCR, CR, VGPR, or PR are defined in outcome measure #4. PD is having any 1 or more of following criteria: increase of 25% from lowest confirmed response value; increase between involved and uninvolved FLC levels >10 mg/dL; increase in BM plasma-cell ≥10%; appearance of new lesion, ≥ 50% increase in sum of products of 2 longest perpendicular diameters of >1 lesion, or ≥ 50% increase in longest diameter of a previous lesion >1 cm in short axis; ≥ 50% increase in circulating plasma cells. Relapse is new soft tissue plasmacytomas or bone lesions; increase in size of existing plasmacytomas or bone lesions; hypercalcemia (> 11 mg/dL); decrease in hemoglobin of ≥ 2 g/dL; rise in serum creatinine by 2 mg/dL; hyperviscosity. Kaplan Meier estimates were used.
Time Frame: Up to 1.5 years
Population: Participants in the Full Analysis Set who had objective response were analyzed. Participants who were observed to have documented relapse, documented PD, or death were censored at the date of their last response assessment.
  As all participants were dosed with same dose of magrolimab, per prespecified analysis, data for Safety Run-in and corresponding Dose-expansion cohorts were combined for all 3 arms.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Magrolimab+Daratumumab | Magrolimab+Pomalidomide+Dexamethasone | Magrolimab+Carfilzomib+Dexamethasone
Number analyzed (Participants) | 2 | 2 | 4
months | NA [NA to NA] — Median, upper and lower limit of confidence interval (CI) were not estimable due to low number of participants with events. | NA [3.9 to NA] — Median and upper limit of CI were not estimable due to low number of participants with events. | NA [NA to NA] — Median, upper and lower limit of CI were not estimable due to low number of participants with events.

6. Secondary Outcome: Serum Concentration of Magrolimab
Description: Arm 1: Magrolimab+Daratumumab; Arm 2: Magrolimab+Pomalidomide+Dexamethasone; Arm 3: Magrolimab+Carfilzomib+Dexamethasone.
Time Frame: Arm 1, 2, 3: Predose: Days 1 and 22 of Cycle 1, Day 1 of Cycles 2, 3, 4, 5, 7, and on last sample collection day (anytime; up to Day 358); Arm 1 and 3: Predose: Day 1 of Cycles 10 and 13
Population: The Pharmacokinetic Analysis Set included all participants who received ≥ 1 dose of magrolimab and had ≥ 1 measurable posttreatment serum concentration of magrolimab. Participants with available data were analyzed.
  As all participants were dosed with same dose of magrolimab, per prespecified analysis, data for Safety Run-in and corresponding Dose-expansion cohorts were combined for all 3 arms.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Magrolimab+Daratumumab | Magrolimab+Pomalidomide+Dexamethasone | Magrolimab+Carfilzomib+Dexamethasone
Number analyzed (Participants) | 10 | 10 | 10
ng/mL
  Predose: Cycle 1 Day 1 | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation | NA (NA) — Mean and standard deviation were not calculable as the values were below the limit of quantitation
  Predose: Cycle 1 Day 22: number analyzed (Participants) | 8 | 8 | 7
  Predose: Cycle 1 Day 22 | 435000 (245000) | 303000 (182000) | 421000 (115000)
  Predose: Cycle 2 Day 1: number analyzed (Participants) | 7 | 5 | 8
  Predose: Cycle 2 Day 1 | 621000 (233000) | 713000 (293000) | 675000 (274000)
  Predose: Cycle 3 Day 1: number analyzed (Participants) | 4 | 6 | 8
  Predose: Cycle 3 Day 1 | 853000 (399000) | 739000 (365000) | 847000 (238000)
  Predose: Cycle 4 Day 1: number analyzed (Participants) | 2 | 1 | 2
  Predose: Cycle 4 Day 1 | 694000 (82700) | 5540 (NA) — Standard deviation was not calculable due to less than 3 participants available for analysis. | 459000 (161000)
  Predose: Cycle 5 Day 1: number analyzed (Participants) | 3 | 5 | 5
  Predose: Cycle 5 Day 1 | 517000 (186000) | 373000 (142000) | 448000 (90700)
  Predose: Cycle 7 Day 1: number analyzed (Participants) | 1 | 3 | 4
  Predose: Cycle 7 Day 1 | 332000 (NA) — Standard deviation was not calculable due to less than 3 participants available for analysis. | 307000 (153000) | 376000 (140000)
  Predose: Cycle 10 Day 1: number analyzed (Participants) | 1 | 0 | 2
  Predose: Cycle 10 Day 1 | 336000 (NA) — Standard deviation was not calculable due to less than 3 participants available for analysis. |  | 361000 (345000)
  Predose: Cycle 13 Day 1: number analyzed (Participants) | 1 | 0 | 1
  Predose: Cycle 13 Day 1 | 295000 (NA) — Standard deviation was not calculable due to less than 3 participants available for analysis. |  | 624000 (NA) — Standard deviation was not calculable due to less than 3 participants available for analysis.
  Anytime: Last sample collection day: Up to Day 358: number analyzed (Participants) | 9 | 6 | 2
  Anytime: Last sample collection day: Up to Day 358 | 445000 (337000) | 179000 (131000) | 86000 (34000)

7. Secondary Outcome: Percentage of Participants With Positive Anti-magrolimab Antibodies
Description: The percentage of participants who had treatment induced or treatment-boosted anti-drug antibody (ADA) based on participants who had non-missing baseline ADA sample and at least one post-treatment ADA result reported in Immunogenicity Analysis Set. Treatment-Induced ADA: participants who had negative baseline ADA sample and at least one positive post-treatment ADA sample based on participants who had both non-missing baseline and at least one post-treatment ADA result reported. Treatment-Boosted ADA: participants who had positive baseline ADA sample and at least one positive post-treatment ADA sample and the (max titer of the posttreatment ADA) / (titer of baseline ADA) >= 4.
Time Frame: Up to Day 358
Population: The Immunogenicity Analysis Set included all enrolled participants who received at least 1 dose of magrolimab and have at least 1 evaluable anti-magrolimab antibody test result.
  As all participants were dosed with same dose of magrolimab, per prespecified analysis, data for Safety Run-in and corresponding Dose-expansion cohorts were combined for all 3 arms.
Measure: Number; unit: percentage of participants
Arm/Group | Magrolimab+Daratumumab | Magrolimab+Pomalidomide+Dexamethasone | Magrolimab+Carfilzomib+Dexamethasone
Number analyzed (Participants) | 10 | 8 | 10
percentage of participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality: Up to 1.5 years; Adverse events: Up to 1.3 years plus 70 days
Description: All-cause mortality: The All Enrolled Analysis Set included all participants who received a study patient identification number in study after screening. Adverse events: The Safety Analysis Set included all participants who received at least 1 dose of study treatment with treatment group designated according to the actual treatment received.
  Per prespecified analysis, data for Safety Run-in and corresponding Dose-expansion cohorts were combined for all 3 arms.
Arm/Group | Magrolimab+Daratumumab | Magrolimab+Pomalidomide+Dexamethasone | Magrolimab+Carfilzomib+Dexamethasone
All-Cause Mortality (participants affected / at risk) | 4/15 | 4/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 5/14 | 5/10 | 4/11
Other Adverse Events (participants affected / at risk) | 14/14 | 10/10 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Magrolimab+Daratumumab (N=14) | Magrolimab+Pomalidomide+Dexamethasone (N=10) | Magrolimab+Carfilzomib+Dexamethasone (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Covid-19 pneumonia (Infections and infestations) | 0 | 1 | 0
Febrile infection (Infections and infestations) | 0 | 1 | 0
Klebsiella urinary tract infection (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 2
Sepsis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Assisted suicide (Surgical and medical procedures) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Magrolimab+Daratumumab (N=14) | Magrolimab+Pomalidomide+Dexamethasone (N=10) | Magrolimab+Carfilzomib+Dexamethasone (N=11)
Anaemia (Blood and lymphatic system disorders) | 7 | 6 | 6
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 2
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 1 | 0
Eye pain (Eye disorders) | 1 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 2 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 0 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 4
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 3 | 3
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1
Asthenia (General disorders) | 1 | 2 | 0
Chills (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 6 | 3 | 6
Gait disturbance (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 1 | 3
Peripheral swelling (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 2 | 1 | 2
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 3
Candida infection (Infections and infestations) | 1 | 0 | 0
Covid-19 (Infections and infestations) | 1 | 0 | 2
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 2
Respiratory tract infection (Infections and infestations) | 1 | 3 | 0
Sinusitis (Infections and infestations) | 1 | 2 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 2 | 2
Viral infection (Infections and infestations) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 3
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 2
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 4 | 0 | 2
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 1
Blood calcium increased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 3 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1
Blood uric acid increased (Investigations) | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 2 | 0
Lymphocyte count decreased (Investigations) | 0 | 2 | 2
Neutrophil count decreased (Investigations) | 2 | 4 | 2
Platelet count decreased (Investigations) | 2 | 3 | 7
Weight decreased (Investigations) | 0 | 1 | 0
White blood cell count decreased (Investigations) | 2 | 2 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Coordination abnormal (Nervous system disorders) | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 2
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 5 | 2 | 3
Paraesthesia (Nervous system disorders) | 1 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1
Device breakage (Product Issues) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 3 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 2 | 2 | 1
Hypotension (Vascular disorders) | 0 | 1 | 1

LIMITATIONS AND CAVEATS:
This study was terminated early due to the Sponsor's decision to discontinue development of the investigational drug and program closure. Due to early termination of the study, reported findings should be interpreted in the context of the study's early closure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/46/NCT04892446/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-13): https://cdn.clinicaltrials.gov/large-docs/46/NCT04892446/SAP_001.pdf